CLINICAL TRIAL: NCT01233726
Title: Effects of a Complete Diet Rich in Monounsaturated Fatty Acids and Slow Absorption Carbohydrate Administration in Critically Ill Patients With Stress Hyperglycemia. Open Study, Blind Randomised, Multicenter and Controlled.
Brief Title: Effects of a Complete Diet in Critically Ill Patients With Stress Hyperglycemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vegenat, S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IR2009; DIABET IR IDI-20080283 (Other: VEGENAT, S.A.)
Record Dates: First submitted 2010-10-29; First posted 2010-11-03 (Estimated); Results first posted 2016-09-01 (Estimated); Last update posted 2016-09-01 (Estimated); Status verified 2016-07

CONDITIONS: Critical Illness; Hyperglycemia; Dietary Modification; Metabolic Stress Hyperglycemia; Mechanical Ventilation Complication
Keywords: Critical illness; Hyperglycemia; Mechanical Ventilation; Enteral nutrition; T-Diet plus Diabet IR; Malnutrition; Insulin resistance; Metabolic stress
MeSH Terms: conditions — Critical Illness; Hyperglycemia; Malnutrition; Insulin Resistance | interventions — Phentermine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- T-DIET PLUS DIABET IR (Experimental): Patients of this group will receive T-Diet plus Diabet IR as unique nutritional support throughout the day, receiving 25 kcal / kg • day (from the first 48 hours after checking tolerance) via gastric or transpyloric
  Interventions: Dietary Supplement: T-Diet plus Diabet IR
- ISOSOURCE PROTEIN FIBRE (Active Comparator): Patients of this group will receive ISOSOURCE PROTEIN FIBRE (Nestlé Nutrition) as unique nutritional support throughout the day receiving 25 kcal / kg • day (from the first 48 hours after checking tolerance) via gastric or transpyloric
  Interventions: Dietary Supplement: ISOSOURCE PROTEIN FIBRE
- GLUCERNA SELECT (Active Comparator): Patients of this group will receive GLUCERNA SELECT (Abbott Laboratories) as unique nutritional support throughout the day, receiving 25 kcal / kg • day (from the first 48 hours after checking tolerance) via gastric or transpyloric
  Interventions: Dietary Supplement: GLUCERNA SELECT

INTERVENTIONS:
Dietary Supplement: T-Diet plus Diabet IR — Group 1 will receive, 25 kcal / kg • day for 28 days, via gastric or transpyloric.
  Other Names: DIABA HP
  Arms: T-DIET PLUS DIABET IR
Dietary Supplement: ISOSOURCE PROTEIN FIBRE — Group 2 will receive, 25 kcal / kg • day for 28 days, via gastric or transpyloric.
  Other Names: ISS PROT FIB
  Arms: ISOSOURCE PROTEIN FIBRE
Dietary Supplement: GLUCERNA SELECT — Group 3 will receive, 25 kcal / kg • day for 28 days, via gastric or transpyloric.
  Other Names: GLUC SEL
  Arms: GLUCERNA SELECT

SUMMARY:
The aim of the study is to evaluate the beneficial effects of the administration of a complete diet rich in monounsaturated fatty acids (MUFA) and slow absorption carbohydrate in patients with stress hyperglycemia(T-Diet Plus Diabet IR).

The main objective of this project is to evaluate blood glucose metabolic control, insulin requirements, insulin action resistance, lipid profile and to reduce infectious complications on mechanical ventilation ICU (intensive care unit) patients after the administration of a complete diet enriched in MUFA and slow absorption carbohydrates, without fructose.

DETAILED DESCRIPTION:
Enteral formula administration designed for critically ill patients in metabolic stress situations, hyperglycemia and insulin resistance, formulated with monounsaturated fatty acids (MUFA), slowly absorption carbohydrates, omega-3 series polyunsaturated fatty acids (PUFA)enriched in eicosapentanoic acid (EPA) and docosahexaenoic acid (DHA), should be associated with an improvement in metabolic control, based on glucose levels reduction, and a decrease of insulin resistance infectious complications , mechanical ventilation days, ICU and hospital stay. All this against other two high protein conventional specific diets for hyperglycaemia patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 admitted to intensive care units (ICU), with mechanical ventilation.
* Patients receiving EN (enteral nutrition), for 5 days or more.
* ICU stay in 48 hours or less, in the time of study inclusion.
* Patients developing hyperglycemia in 48 hours of stay in ICU.
* Nutritional support initiation within 48 hours of stay in ICU.

Exclusion Criteria:

* Patients with a life expectancy less than 48 hours.
* Patients participating in another study.
* Patients with APACHE II (Acute Physiology and Chronic Health Evaluation) less than 10.
* Patients with BMI (body mass index) > 40 Kg/m2.
* Patients with Type I Diabetes.
* Patients on chronic treatment with corticosteroid dose above 1 mg / kg / day of methylprednisolone or equivalent.
* Pregnant patients.
* Patients taking lipid-lowering drugs.
* Acute renal failure patients, defined by the following criteria:

  * Serum creatinine greater than 4 mg / dL with acute rise higher than 0.5 mg / dl / day.
  * Serum creatinine higher than 3 mg/dL.
  * Diuresis < 0.3 ml/kg/h during 24 hours.
  * Anury for 12 hours or more.
* Hepatic failure patients, defined by the following parameters:

  * Serious acute hepatic failure.
  * Child degrees B-C.
  * Serum bilirubin higher than 3 mg/dL.
* Patients with parenteral nutrition during study inclusion.
* Informed consent absence.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2010-04; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alfonso Mesejo, PhD, Principal Investigator — Hospital Clinico Universitario de Valencia; Juan Carlos Montejo, PhD, Principal Investigator — Hospital Universitario 12 de Octubre
Locations (2):
- Spain (2):
  - Intensive Care Unit. Hospital Universitario 12 de Octubre, Madrid, Madrid
  - Intensive Care Unit. Hospital Clinico Universitario de Valencia, Valencia, Valencia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mesejo A, Montejo-Gonzalez JC, Vaquerizo-Alonso C, Lobo-Tamer G, Zabarte-Martinez M, Herrero-Meseguer JI, Acosta-Escribano J, Blesa-Malpica A, Martinez-Lozano F. Diabetes-specific enteral nutrition formula in hyperglycemic, mechanically ventilated, critically ill patients: a prospective, open-label, blind-randomized, multicenter study. Crit Care. 2015 Nov 9;19:390. doi: 10.1186/s13054-015-1108-1. PMID 26549276

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study examines whether a high-protein diabetes-specific formula reduces insulin needs, improves glycemic control and reduces ICU-adquired infection in critically ill, hyperglycemic patients on mechanical ventilation (MV)
Pre-assignment Details: The study was performed over the period April 2010 to May 2012. A website was constructed to record data and to randoize patients to each EN formula. Data were collected online using an electronic case report form.
Groups:
- DIABA HP: Patients of this group received Diaba HP as unique nutritional support throughout the day, receiving 25 kcal / kg /day (from the first 48 hours after checking tolerance) via gastric or transpyloric
  Diaba HP: Diaba HP is a complete normocaloric high protein diet, indicated for the dietary management of diabetic patients or hyperglycemia related malnutrition.
  DIABA HP group received, 25 kcal / kg /day for 28 days, via gastric or transpyloric.
- ISOSOURCE PROTEIN FIBRE: Patients of this group received ISOSOURCE PROTEIN FIBRE (Nestlé Nutrition) as unique nutritional support throughout the day, receiving 25 kcal / kg /day (from the first 48 hours after checking tolerance) via gastric or transpyloric
  ISOSOURCE PROTEIN FIBRE: Isosource protein fibre is a complete high protein diet with fibre mixture.
  ISOSOURCE PROTEIN FIBRE group received, 25 kcal / kg / day for 28 days, via gastric or transpyloric.
- GLUCERNA SELECT: Patients of this group received GLUCERNA SELECT (Abbott Laboratories) as unique nutritional support throughout the day, receiving 25 kcal / kg /day (from the first 48 hours after checking tolerance) via gastric or transpyloric
  GLUCERNA SELECT: Glucerna Select is a complete high protein special formula, with fiber, enriched in monounsaturated fatty acids, with slow absorption carbohydrates.
  GLUCERNA SELECT group will received 25 kcal / kg / day for 28 days, via gastric or transpyloric.
Period: Overall Study
Arm/Group | DIABA HP | ISOSOURCE PROTEIN FIBRE | GLUCERNA SELECT
Started | 53 | 53 | 53
Completed | 52 | 53 | 52
Not Completed | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Age ≥18 years, ICU stay ≤48 hours upon randomization to EN formula, mechanical ventilation, EN indicated for an expected time ≥5 days. Patients were also required to meet American Diabetes Association criteria for diabetes/hyperglycemia (baseline blood glucose >126 mg/dL after fasting or>200 mg/dL otherwise) in the first 48 h of ICU admission.
Groups:
- DIABA HP: Patients of this group received new-generation diabetes-specific high-protein formula (Diaba HP®, Vegenat, Badajoz, Spain); as unique nutritional support throughout the day, receiving 25 kcal / kg / day (from the first 48 hours after checking tolerance) via gastric or transpyloric
  Diaba HP: Diaba HP is a complete normocaloric high protein diet, indicated for the dietary management of diabetic patients or hyperglycemia related malnutrition.
  DIABA HP group received, 25 kcal / kg/ day for 28 days, via gastric or transpyloric.
- ISOSOURCE PROTEIN FIBRE: Patients of this group will received ISOSOURCE PROTEIN FIBRE (Nestlé Health Science, barcelona, Spain) as unique nutritional support throughout the day, receiving 25 kcal / kg /day (from the first 48 hours after checking tolerance) via gastric or transpyloric
  ISOSOURCE PROTEIN FIBRE: Isosource protein fibre is a complete high protein diet with fibre mixture.
  ISOSOURCE PROTEIN FIBRE group received, 25 kcal / kg / day for 28 days, via gastric or transpyloric.
- GLUCERNA SELECT: Patients of this group will receive GLUCERNA SELECT (Abbott Nutrition, Madrid, Spain) as unique nutritional support throughout the day, receiving 25 kcal / kg / day (from the first 48 hours after checking tolerance) via gastric or transpyloric
  GLUCERNA SELECT: Glucerna Select is a complete high protein special formula, with fiber, enriched in monounsaturated fatty acids, with slow absorption carbohydrates.
  GLUCERNA SELECT group received 25 kcal / kg / day for 28 days, via gastric or transpyloric.
- Total: Total of all reporting groups
Arm/Group | DIABA HP | ISOSOURCE PROTEIN FIBRE | GLUCERNA SELECT | Total
Number analyzed (Participants) | 52 | 53 | 52 | 157
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 57 [43 to 70] | 60 [45 to 71] | 58 [46 to 68] | 58 [43 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 10 | 13 | 38
  Male | 37 | 43 | 39 | 119
Body Mass Index (BMI) [Median (Inter-Quartile Range); unit: kg/m^2] | 26 [24 to 29] | 26 [24 to 28] | 26 [24 to 27] | 26 [24 to 29]
APACHE II [Median (Inter-Quartile Range); unit: units on a scale] — Acute Physiology and Chronic Health Evaluation II
  Scale: 0 to 71: based on several measures: at higher score, more severe illness and greater risk of death.
  units on a scale | 17 [14 to 23] | 19 [15 to 22] | 19 [16 to 23] | 19 [14 to 23]
SOFA score [Median (Inter-Quartile Range); unit: units on a scale] — Sepsis-related Organ Failure Assessment score.
  Score:
  0-6: 10% of mortality; 7-9: 15-20% of mortality; 10-12: 40-50% of mortality; 13-14: 50-60 % of mortality; 15: >80% of mortality; 16-24: >90% of mortality.
  units on a scale | 8 [6 to 14] | 7 [5 to 12] | 7 [4 to 12] | 8 [4 to 14]
Calorie requirements [Geometric Mean (Standard Deviation); unit: kcal/day] | 1690.4 (384.9) | 1707.1 (275.4) | 1728.2 (309.2) | 1708.6 (323.2)
Start of EN [Median (Inter-Quartile Range); unit: hours] — Start of Enteral Nutrition: elapsed time from admission to start enteral nutrition
  hours | 23.4 [18.1 to 27.2] | 25.1 [19.6 to 26.2] | 26.7 [21.3 to 28] | 25.1 [18.1 to 28]
Noninsulin-dependent diabetes [Number; unit: participants] | 11 | 7 | 12 | 30
HbA1c [Mean (Standard Deviation); unit: percentaje of glycated hemoglobin] | 6.34 (1.38) | 5.76 (0.95) | 6.07 (1.39) | 6.1 (1.24)
Capillary glucose level [Mean (Standard Deviation); unit: mg/dL] — Measured after fasting and without insulin infusion for at least 8 hours
  mg/dL | 148.8 (38.8) | 149.9 (38.9) | 151.5 (39.23) | 150 (38.98)
Plasma glucose level [Mean (Standard Deviation); unit: mg/dL] — Measured after fasting and without insulin infusion for at least 8 hours
  mg/dL | 152.1 (54.6) | 147.01 (55.93) | 152.1 (57.12) | 150.4 (55.88)
Insulinemia [Mean (Standard Deviation); unit: microU/mL] — Measured after fasting and without insulin infusion for at least 8 hours
  microU/mL | 21.59 (36.06) | 17.39 (23.77) | 19.15 (20.5) | 19.38 (26.78)
C-peptide [Mean (Standard Deviation); unit: ng/mL] — Measured after fasting and without insulin infusion for at least 8 hours
  ng/mL | 4.61 (3.24) | 4.49 (2.92) | 4.27 (3.67) | 4.46 (3.28)
HOMA2 IR [Mean (Standard Deviation); unit: units on a scale] — HOMA 2: Homeostasis Model Assessment IR: Insulin Resistance. Homeostatic model assessment (HOMA) is a method for assessing β-cell function and insulin resistance (IR) from basal (fasting) glucose and insulin or C-peptide concentrations.
  The HOMA model compares favorably with other models and has the advantage of requiring only a single plasma sample assayed for insulin and glucose. Higher values represent higher insulinemia.
  units on a scale | 2.94 (4.19) | 2.48 (2.76) | 3.38 (2.37) | 2.93 (3.11)
HOMA2 %B [Mean (Standard Deviation); unit: % of beta cell function] — HOMA 2: Homeostasis Model Assessment B: Beta cell function.
  Homeostatic model assessment (HOMA) is a method for assessing β-cell function and insulin resistance (IR) from basal (fasting) glucose and insulin or C-peptide concentrations.
  % of beta cell function | 102.6 (57.81) | 110.5 (74.34) | 96.55 (85.09) | 103.21 (72.41)
HOMA2 %S [Mean (Standard Deviation); unit: % of insulin sensitivity] — HOMA2: Homeostasis Model Assessment S: Insulin Sensitivity
  % of insulin sensitivity | 79.12 (75.2) | 69.6 (48.7) | 68.09 (66.9) | 72.27 (63.6)
Infection [Number; unit: participants] — Number of patients with infection from any source
  participants | 13 | 15 | 8 | 36
Diagnostic group: Medical [Number; unit: participants] | 32 | 36 | 30 | 98
Diagnostic group: Trauma [Number; unit: participants] | 13 | 9 | 15 | 37
Diagnostic group: Surgery [Number; unit: participants] | 7 | 8 | 7 | 22

OUTCOME MEASURES:

1. Primary Outcome: Measure of Biochemical Parameters and Evaluation of Infectious Complications 1
Description: The variables recorded related to glycemic control in mg/dL are provided in this table.
Time Frame: 28 days post-admission
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- Diaba HP: Patients of this group received Diaba HP as unique nutritional support throughout the day, receiving 25 kcal / kg /day (from the first 48 hours after checking tolerance) via gastric or transpyloric
  Diaba HP: Diaba HP is a complete normocaloric high protein diet, indicated for the dietary management of diabetic patients or hyperglycemia related malnutrition.
  Group Diaba HP received, 25 kcal / kg /day for 28 days
- ISOSOURCE PROTEIN FIBRE: Patients of this group will receive ISOSOURCE PROTEIN FIBRE (Nestlé Nutrition) as unique nutritional support throughout the day, receiving 25 kcal / kg • day (from the first 48 hours after checking tolerance) via gastric or transpyloric
  ISOSOURCE PROTEIN FIBRE: Isosource protein fibre is a complete high protein diet with fibre mixture.
  Group Isosource protein fibre will receive, 25 kcal / kg • day for 28 days, via gastric or transpyloric.
- GLUCERNA SELECT: Patients of this group will receive GLUCERNA SELECT (Abbott Laboratories) as unique nutritional support throughout the day, receiving 25 kcal / kg • day (from the first 48 hours after checking tolerance) via gastric or transpyloric
  GLUCERNA SELECT: Glucerna Select is a complete high protein special formula, with fiber, enriched in monounsaturated fatty acids, with slow absorption carbohydrates.
  Group GLUCERNA SELECT will receive 25 kcal / kg • day for 28 days, via gastric or transpyloric.
Arm/Group | Diaba HP | ISOSOURCE PROTEIN FIBRE | GLUCERNA SELECT
Number analyzed (Participants) | 52 | 53 | 52
mg/dL
  Plasma glucose level (mg/dL) | 138.6 (39.1) | 146.1 (49.9) | 143.9 (45.9)
  Capillary glucose level (mg/dL) | 146.1 (45.8) | 155.3 (63.6) | 150.1 (41.9)
  Mean capillary glycemia on ICU day 1 (mg/dL) | 147.5 (40.2) | 160 (55.5) | 145.6 (46.6)
  Peak glucose level (mg/dL) | 181.3 (52) | 193.6 (74.6) | 191.3 (65.8)
  Glycemic variability SD (mg/dL) (ICU days 1-28) | 33.6 (18.4) | 49.1 (21.5) | 41.1 (9.3)
  Glycemic variability SD (mg/dL) (ICU days 1-7) | 43.2 (4.9) | 68.5 (13.5) | 42.5 (2.7)

2. Primary Outcome: Measure of Biochemical Parameters and Evaluation of Infectious Complications 2
Description: The variables recorded related to administered insulin in IU/day are provided in this table
Time Frame: 28 days post-admission
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: IU/day
Arm/Group | Diaba HP | ISOSOURCE PROTEIN FIBRE | GLUCERNA SELECT
Number analyzed (Participants) | 52 | 53 | 52
IU/day | 19.1 (13.1) | 23.7 (40.1) | 20.3 (30.1)

3. Primary Outcome: Measure of Biochemical Parameters and Evaluation of Infectious Complications 3
Description: The variables recorded related to number of capillary glycemia measurements are provided in this table
Time Frame: 28 days post-admission
Population: as for baseline characteristics
Measure: Number; unit: Capillary glycemia measurements
Arm/Group | Diaba HP | ISOSOURCE PROTEIN FIBRE | GLUCERNA SELECT
Number analyzed (Participants) | 52 | 53 | 52
Capillary glycemia measurements | 3605 | 3523 | 3557

4. Primary Outcome: Measure of Biochemical Parameters and Evaluation of Infectious Complications 4
Description: The variables recorded related to the number of measurements per patient per day are provided in this table
Time Frame: 28 days post-admission
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Measurements per patient/day
Arm/Group | Diaba HP | ISOSOURCE PROTEIN FIBRE | GLUCERNA SELECT
Number analyzed (Participants) | 52 | 53 | 52
Measurements per patient/day | 5.7 (3.4) | 5.81 (3.2) | 5.46 (2.9)

5. Primary Outcome: Measure of Biochemical Parameters and Evaluation of Infectious Complications 5
Description: The variables recorded related to Glycemic CV (%) are provided in this table:
  * Glycemic Coeficient of variation (%) after 28 days in ICU
  * Glycemic Coeficient of variation (%) after 7 days in ICU.
Time Frame: 28 days post-admission
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: percentage of Glycemic CV
Arm/Group | Diaba HP | ISOSOURCE PROTEIN FIBRE | GLUCERNA SELECT
Number analyzed (Participants) | 52 | 53 | 52
percentage of Glycemic CV
  Glycemic CV (%) (ICU days 1-28) | 27.9 (5.8) | 32.4 (11.2) | 27.8 (5.2)
  Glycemic CV (%) (ICU days 1-7) | 28.3 (1.9) | 42.6 (8.2) | 28.4 (2.1)

6. Primary Outcome: Primary Outcome: Measure of Biochemical Parameters and Evaluation of Infectious Complications 6.1
Description: This table shows the number of capillary glycemia measurements
Time Frame: 28 days post-admission
Measure: Number; unit: number of capillary glycemia measurement
Arm/Group | Diaba HP | ISOSOURCE PROTEIN FIBRE | GLUCERNA SELECT
Number analyzed (Participants) | 52 | 53 | 52
number of capillary glycemia measurement | 3605 | 3523 | 3557

7. Primary Outcome: Measure of Biochemical Parameters and Evaluation of Infectious Complications 6.2
Description: This table shows the rates of:
  * Controls analysis on 80-150 mg/dL: optimal level of glycemia rate.
  * Hypoglycemia (50-80 mg/dL): moderate hypoglycemia rate.
  * Hypoglycemia (<50 mg/dL): severe hypoglycemia episodes rate.
Time Frame: 28 days post-admission
Population: as for baseline characteristics
Measure: Number; unit: % of capillary glycemia measurements
Arm/Group | Diaba HP | ISOSOURCE PROTEIN FIBRE | GLUCERNA SELECT
Number analyzed (Participants) | 52 | 53 | 52
% of capillary glycemia measurements
  Controls on 80-150 mg/dL | 59 | 57.6 | 59.59
  Hypoglycemia (50-80 mg/dL) | 1.48 | 3.63 | 1.25
  Hypoglycemia (<50 mg/dL) | 0 | 0.11 | 0.02

8. Secondary Outcome: Assessment of Critical Ill Patients Progress During Hospital Stay 1
Description: Infectious complication incidence rate per 100 days of treatment are provided in this table.
Time Frame: 100 days of treatment
Population: as for baseline characteristics
Measure: Number; unit: percentage of patients with infection
Groups:
- ISOSOURCE PROTEIN FIBRE: Patients of this group will receive ISOSOURCE PROTEIN FIBRE (Nestlé Nutrition) as unique nutritional support throughout the day, receiving 25 kcal / kg • day (from the first 48 hours after checking tolerance) via gastric or transpyloric
  ISOSOURCE PROTEIN FIBRE: Isosource protein fibre is a complete high protein diet with fibre mixture.
  ISOSOURCE PROTEIN FIBRE group will receive, 25 kcal / kg • day for 28 days, via gastric or transpyloric.
- GLUCERNA SELECT: Patients of this group will receive GLUCERNA SELECT (Abbott Laboratories) as unique nutritional support throughout the day, receiving 25 kcal / kg • day (from the first 48 hours after checking tolerance) via gastric or transpyloric
  GLUCERNA SELECT: Glucerna Select is a complete high protein special formula, with fiber, enriched in monounsaturated fatty acids, with slow absorption carbohydrates.
  GLUCERNA SELECT group will receive 25 kcal / kg • day for 28 days, via gastric or transpyloric.
Arm/Group | DIABA HP | ISOSOURCE PROTEIN FIBRE | GLUCERNA SELECT
Number analyzed (Participants) | 52 | 53 | 52
percentage of patients with infection | 22 | 24 | 24

9. Secondary Outcome: Assessment of Critical Ill Patients Progress During Hospital Stay 2
Description: Number of participants with catheter-associated bloodstream infection, primary bloodstream infection or urinary tract infection are provided in this table
Time Frame: 28 days post-admission
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | DIABA HP | ISOSOURCE PROTEIN FIBRE | GLUCERNA SELECT
Number analyzed (Participants) | 52 | 53 | 52
participants
  Catether-related bloodstream infection | 1 | 1 | 2
  Primary bloodstream infection | 3 | 1 | 3
  Urinary tract infection | 1 | 1 | 1

10. Secondary Outcome: Assessment of Critical Ill Patients Progress During Hospital Stay 3
Description: The incidence of tracheobronchitis and ventilator-associated pneumonia per 1000 days of mechanical ventilation are provided in this table.
Time Frame: 28 days post-admission
Population: as for baseline characteristics
Measure: Number; unit: number of new cases per 1000 days
Arm/Group | DIABA HP | ISOSOURCE PROTEIN FIBRE | GLUCERNA SELECT
Number analyzed (Participants) | 52 | 53 | 52
number of new cases per 1000 days
  Tracheobonchitis incidence rate | 7 | 10 | 7
  Ventilator-associated pneumonia | 8 | 10 | 6

11. Secondary Outcome: Assessment of Critical Ill Patients Progress During Hospital Stay 4
Description: Number of participants with infectious complications is provided in this table.
Time Frame: 100 days of treatment
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Diaba HP | ISOSOURCE PROTEIN FIBRE | GLUCERNA SELECT
Number analyzed (Participants) | 52 | 53 | 52
participants | 18 | 23 | 23

ADVERSE EVENTS:
Time Frame: All participants were followed at the ICU for a maximum of 28 days.
Description: No adverse effects have been observed and/or registered related with the products intake during the clinical trial period. Data provided in outcome measure are related with the individual patology of each patient, not with the product intake (enteral nutrition intake).
Groups:
- DIABA HP: Patients of this group received Diaba HP® as unique nutritional support throughout the day, receiving 25 kcal / kg / day (from the first 48 hours after checking tolerance) via gastric or transpyloric
  Diaba HP is a complete normocaloric high protein diet, indicated for the dietary management of diabetic patients or hyperglycemia related malnutrition.
  DIABA HP group received, 25 kcal / kg /day for 28 days, via gastric or transpyloric.
- ISOSOURCE PROTEIN FIBRE: Patients of this group will receive ISOSOURCE PROTEIN FIBRE (Nestlé Nutrition) as unique nutritional support throughout the day, receiving 25 kcal / kg / day (from the first 48 hours after checking tolerance) via gastric or transpyloric
  ISOSOURCE PROTEIN FIBRE: Isosource protein fibre is a complete high protein diet with fibre mixture.
  ISOSOURCE PROTEIN FIBRE group received, 25 kcal / kg / day for 28 days, via gastric or transpyloric.
- GLUCERNA SELECT: Patients of this group will receive GLUCERNA SELECT (Abbott Laboratories) as unique nutritional support throughout the day, receiving 25 kcal / kg/ day (from the first 48 hours after checking tolerance) via gastric or transpyloric
  GLUCERNA SELECT: Glucerna Select is a complete high protein special formula, with fiber, enriched in monounsaturated fatty acids, with slow absorption carbohydrates.
  GLUCERNA SELECT group will receive 25 kcal / kg / day for 28 days, via gastric or transpyloric.
Arm/Group | DIABA HP | ISOSOURCE PROTEIN FIBRE | GLUCERNA SELECT
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/53 | 0/52
Other Adverse Events (participants affected / at risk) | 0/52 | 0/53 | 0/52

LIMITATIONS AND CAVEATS:
No overall limitations and caveats have been observed and/or registered related with the products intake during the clinical trial period.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes